CLINICAL TRIAL: NCT06535906
Title: Effect of Manual Lymphatic Drainage and Kinesio Taping on Delayed Onset Muscle Soreness: Randomized -Controlled Study
Brief Title: Effect of Manual Lymphatic Drainage and Kinesio Taping on Delayed Onset Muscle Soreness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Yavuz Özkan, Master Student Physiotherapist, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEU-FTR-YO-01
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Delayed Onset Muscle Soreness
Keywords: delayed onset muscle soreness; kinesio taping; manual lymphatic drainage; pressure pain threshold; pain
MeSH Terms: conditions — Pain | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Intervention Model Description: We conducted our study as a randomized controlled study. There will be no masking in our study.
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- kinesio taping (Active Comparator): Kinesio taping is a widely used physiotherapy application for muscle pain. Kinesio taping will be applied to patients in this group.
  Interventions: Other: kinesio taping
- placebo kinesio taping (Placebo Comparator): Kinesio taping is a widely used physiotherapy application for muscle pain. In this group, placebo kinesio taping will be applied to the patients.
  Interventions: Other: placebo kinesio taping
- manual lymph drainage (Active Comparator): Manual lymphatic drainage is a method commonly used in cases where lymph flow is impaired. Manual lymphatic drainage will be applied to patients in this group.
  Interventions: Other: manual lymph drainage
- placebo manual lymph drainage (Placebo Comparator): Manual lymphatic drainage is a method commonly used in cases where lymph flow is impaired. In this group, patients will receive placebo manual lymphatic drainage.
  Interventions: Other: placebo manual lymph drainage

INTERVENTIONS:
Other: kinesio taping — The 5 cm wide Kinesio tape (Kinesio® Tex Gold™, Albuquerque, NM) applied to the participants has the ability to stretch up to 140% of its original length. Moreover, it provides comfortable use for 3 to 5 days thanks to its latex-free, cotton, hypoallergenic and porous features. The skin will be cleaned with alcohol before applying Kinesio tape. To prevent muscle tension, the physiotherapist will apply the kinesio tape inhibition technique to the wrist flexor muscles with light tension (15-25% of the current tension) from the end point to the origin. We will use this inhibition technique to prevent muscle spasm. Kinesio taping will be applied immediately after exercise
  Arms: kinesio taping
Other: placebo kinesio taping — 5 cm wide and 0.5 mm thick I-shaped Kinesio tape (Kinesio Tex® Gold) will be used. The tape will be applied in a plus-shaped, tension-free and technical sitting position. Kinesio taping will be applied immediately after exercise
  Arms: placebo kinesio taping
Other: manual lymph drainage — Participants will lie in a supine position with their knees bent. Manual lymphatic drainage will begin with abdominal lymph drainage followed by central lymph stimulation. Then, bilateral axillary lymph nodes will be stimulated and the fluid in the exercised arm will be directed to the axillary lymph nodes. While the patients are in the prone position, the axillary lymph nodes will be stimulated in the same way and each manual lymphatic drainage will be performed from the back to the axillary lymph node. Each treatment session will last approximately 30 minutes
  Arms: manual lymph drainage
Other: placebo manual lymph drainage — Participants will lie in a supine position with their knees bent. It will only be moved in a stroking style with hand contact from the fingers towards the armpit.
  Arms: placebo manual lymph drainage

SUMMARY:
Delayed muscle soreness is pain and tenderness that occurs after unusual exercises, most often involving eccentric contraction. This sensitivity, which usually begins in the distal part of the muscle and is intense, spreads progressively throughout the entire muscle 24-48 hours after exercise. The intensity of the discomfort increases within the first 24 hours following cessation of exercise, peaks between 24 and 72 hours, decreases and eventually disappears within 5-7 days after exercise.

Delayed onset muscle soreness is considered one of the most common and recurring forms of sports injuries. The most prominent symptoms and findings are a decrease in joint range of motion and strength, edema, stiffness, pain and tenderness. In the planned study, the investigatorss aimed to compare the effects of kinesio taping, manual drainage, placebo kinesio taping and placebo kinesio taping on pain intensity, pain threshold and tolerance, sensory sensitivity and connective tissue stiffness in individuals with delayed-onset muscle soreness.48 healthy adults will be included in our study. Participants will be divided into four groups of 12 people: kinesio taping, placebo kinesio taping, manual lymph drainage and placebo manual lymph drainage. Our participants will have a maximum repetition weight on their wrist flexor muscles, and a delayed muscle soreness protocol will be applied using 80% of this amount. In our participants, pain at rest and activity (VAS), pressure pain threshold and tolerance (algometer), tactile sense (Semmes-Weinstein Monofilament Test), edema (circumference measurement with tape measure), treatment satisfaction and effect (VAS), tissue tension (skin rolling). and perceived fatigue (VAS) will be evaluated. The researchers plan to conduct 5 assessments: before the delayed-onset muscle soreness protocol, immediately after the protocol, immediately after treatment, and 24 hours and 48 hours after the initial assessment.

DETAILED DESCRIPTION:
Volunteers, healthcare students and university employees between the ages of 18-40 who meet the inclusion criteria will be included in our study. All participants meeting the inclusion criteria will be selected and divided into four groups using computer-generated randomization (simple randomization) ( www.randomizer.org ).Participants will be divided into four groups: manual lymph drainage, placebo manual lymph drainage, kinesio taping and placebo kinesio taping.

On the first day, after the volunteers who meet the inclusion criteria are divided into groups, demographic information (gender, age, height, body weight) will be collected. The first evaluation will be made after demographic information is obtained. The evaluation includes pain at rest and activity (VAS), pressure pain threshold and tolerance (algometer), tactile sense (Semmes-Weinstein Monofilament Test), edema (circumference measurement with tape measure), treatment satisfaction and effect (VAS), tissue tension and perceived fatigue. (VAS) will be evaluated. Visual Analog scale will be used to evaluate pain at rest and activity. Visual Analog Scale is a 10 cm long ruler drawn horizontally, starting with "No pain" and ending with "Unbearable pain". Our participants will be asked to mark an "x" in the appropriate area on this ruler for the intensity of pain they feel at rest. In order to determine the intensity of pain during the activity, the patient will be asked to perform wrist flexion and extension and will be asked to mark the pain they feel during the movement on the ruler in the same way. Algometer will be used to evaluate pressure pain threshold and tolerance. As the measurement point, the researcher will mark 5 cm distal to the medial epicondyle of the humerus on the line connecting the midpoint of the wrist joint and the medial epicondyle of the humerus . Two measurements will be made on this point with an interval of 30 seconds and the average will be recorded. Semmes-Weinstein Monofilament Test will be used for tactile sensation. The patient is asked to close his eyes while sitting with his forearm supported. The point where the pressure pain threshold was measured was chosen as the measurement point. Monofilament test is applied to the determined area a maximum of 3 times; Force is applied until the filament becomes slightly curved. The participant is told to say yes as soon as he feels it and the application is stopped at that moment. For each filament that is not felt, the next value, the thicker filament, is tried. Each filament is kept in the applied area for 1-1.5 seconds. The value obtained after the measurement is recorded. Edema measurement will be measured with a non-flexible tape measure at the reference point where the pressure pain threshold is measured, with the participant in a sitting position with forearm supported. Treatment satisfaction and impact will only be questioned at the final evaluation.Researchers will evaluate the patient's treatment satisfaction level with a visual analog scale. The patient will be asked to evaluate his/her satisfaction with the treatment by placing an "x" mark on the ruler, which starts with "I am not at all satisfied" and ends with "I am very satisfied". Tissue tension will be evaluated on the forearm with the skin rolling technique. Visual Analog scale will be used for perceived fatigue. "There is no fatigue at all." The patient will be asked to evaluate the fatigue he/she feels by placing an "x" on the ruler starting with "Severe Fatigue". All evaluations will be applied to the non-dominant upper extremity wrist flexor muscles. Because the researchers recruited healthy volunteers, they do not expect the participants to experience any pain at the start of the study.Researchers will create the muscle soreness they want using free weights. Researchers will find a 1 Maximum Rep Weight to create delayed onset muscle soreness. Researchers will reference previous studies to find a 1 Maximum Rep Weight.1 Maximum Repetition is the weight that can be lifted only once but cannot be lifted a second time. 1 After the Maximum Repetition weight is determined, an eccentric exercise program will be applied to the participants with a free weight of 80% of this weight. After the first evaluation, the 1 Maximum Repetition weight of the non-dominant wrist flexor muscles will be determined. 1 Mayhew et al.'s formula will be used to find Maximum Repetition. Participants will be given an estimated weight for their wrist flexors and counted the number of times they lift that weight. The resulting weight and number of repetitions will be substituted into the formula and 1 Maximum Repetition will be calculated. After 1 Maximum Repetition is determined, a delayed muscle soreness protocol will be applied by performing 10 sets of wrist flexion consisting of 10 repetitions at 80% of 1 Maximum Repetition. There will be a 1 minute rest period between each set. After delayed onset muscle soreness is established, participants will be given a second evaluation and then their treatments will be applied according to the groups they belong to. After the treatment, the third evaluation will be made and the first day applications will end. A fourth assessment will be made 24 hours after the delayed muscle soreness protocol and a fifth assessment will be made 48 hours later.All of the parameters described above will be evaluated in all five planned evaluations. Treatment satisfaction and impact will only be questioned at the final evaluation

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-40
* Agreeing to participate in the study
* Being healthy sedentary

Exclusion Criteria:

* Those with neurological or perception problems
* Having any musculoskeletal injury in the last 6 months
* Having pain in the upper extremity and a history of surgery
* Participating in upper extremity weight training in the last 6 months
* Those taking anti-inflammatory or analgesic medications up to 12 hours before evaluation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Pain at rest and activity | Three days
  It will be evaluated with a visual analog scale. Possible scores range from 0 (no pain) to 10 (worst possible pain)
Pressure pain threshold and tolerance | Three days
  It will be measured with an algometer. The result will be displayed in pounds

SECONDARY OUTCOMES:
Tactile sensation | Three days
  Semmes-Weinstein Monofilament Test will be used for tactile sensation.Monofilament sets containing sizes 2.83, 3.61, 4.31, 4.56, 6.65 will be used.
Edema | Three days
  Edema measurement will be made with a non-flexible tape measure. Will be recorded in centimeters
Tissue tension | Three days
  Tissue tension will be evaluated on the forearm with the skin rolling technique. In all planned evaluations, the tension bands will be evaluated according to the amount of tension (sensitivity) felt by the individual and the amount of tension felt by the therapist as "none (0)", "mild (1)", "moderate (2)" and "severe (3)".
Treatment satisfaction and impact | One day
  It will be evaluated with a visual analog scale. It will be scored between 0 - 10. 0(I am not happy at all)- 10(I am completely satisfied)
perceived fatigue | Three days
  It will be evaluated with a visual analog scale. It will be scored between 0 - 10. 0(I'm not tired at all) - 10(I'm completely tired).

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Özkan, MSc, Principal Investigator — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No